CLINICAL TRIAL: NCT00052338
Title: A Phase I Study Of PS-341 In Combination With Gemcitabine And Carbloplatin In Selected Stage IIIB Or IV Non-Small Cell Lung Cancer
Brief Title: Bortezomib Plus Gemcitabine and Carboplatin in Treating Patients With Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02503; PHI-40; N01CM17101 (NIH); CDR0000258189 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Pleural Effusion; Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin; Bortezomib

ARMS (1):
- Treatment (gemcitabine hydrochloride, carboplatin, bortezomib) (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8, carboplatin IV over 15-30 minutes on day 1, followed 1 hour later by bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with a clinical or radiographic response may continue receiving bortezomib beyond 6 courses.
  Interventions: Drug: gemcitabine hydrochloride; Drug: carboplatin; Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug and bortezomib may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of combining bortezomib with gemcitabine and carboplatin in patients with advanced or recurrent non-small cell lung cancer.

II. Determine the maximum tolerated dose of bortezomib administered in combination with gemcitabine and carboplatin in these patients.

III. Correlate results from laboratory studies on patient tissue and serum specimens with potential predictors of response in patients treated with this regimen.

IV. Determine, preliminarily, the response of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8, carboplatin IV over 15-30 minutes on day 1, followed 1 hour later by bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with a clinical or radiographic response may continue receiving bortezomib beyond 6 courses.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, at least 10 additional patients with chemotherapy-naive disease receive treatment as above with the MTD of bortezomib.

Patients are followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Selected stage IIIB (malignant pleural effusion) or stage IV disease
  * Recurrent disease after first-line therapy allowed
* Patients who received prior platinum-based chemotherapy must have no disease progression during or within 3 months after completion of therapy

  * Patients who are enrolled at the maximum tolerated dose must have chemotherapy-naïve disease
* Evaluable disease
* Asymptomatic brain metastases allowed if treated with surgical resection or radiotherapy, neurologically stable, and off steroids for at least 4 weeks
* Performance status - Karnofsky 60-100%
* More than 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 50 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy grade 2 or greater
* No prior allergic reactions to compounds of similar chemical or biological composition to bortezomib or other agents used in this study
* No concurrent ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No concurrent routine filgrastim (G-CSF)
* See Disease Characteristics
* No more than 1 prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* No prior gemcitabine
* See Disease Characteristics
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* See Disease Characteristics
* More than 30 days since prior investigational drugs
* No prior bortezomib
* No concurrent anticonvulsant therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies with intent to treat malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2002-09; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Toxicities at each dose level, graded using the CTC version 2.0 | 18 weeks
  Summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity, (by NCI Common Toxicity Criteria and nadir or maximum values for the laboratory measures, time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and course.

SECONDARY OUTCOMES:
Response rate, assessed by standard RECIST criteria | Up to 2 years
  Summarized by exact binomial confidence intervals.
Survival | From registration to time of death due to any cause, assessed up to 2 years
  Summarized with Kaplan-Meier plots.
Time to failure | Up to 2 years
  Summarized with Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Davies, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States